CLINICAL TRIAL: NCT02373007
Title: Evaluation of Safety and Effectiveness Modified Scopinaro Technique in the Surgical Treatment of Obesity Compared to Classical Scopinaro Technique
Brief Title: Evaluation of Two Surgical Scopinaro Techniques in the Treatment of Obesity
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Paulo Reis (Other)
Responsible Party: Principal Investigator, Paulo Reis Esselin de Melo, Paulo Reis Esselin de Melo, Instituto Paulo Reis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTN U1111-1166-7218
Record Dates: First submitted 2015-02-05; First posted 2015-02-26 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Classic Scopinaro Surgery (Other): Patients will get the Bariatric surgery using the Classic Scopinaro Techniques
  Interventions: Procedure: Scopinaro Surgery
- Modified Scopinaro Surgery (Other): Patients will get Bariatric surgery using the Modified Scopinaro Techniques
  Interventions: Procedure: Scopinaro Surgery

INTERVENTIONS:
Procedure: Scopinaro Surgery — Classic Scopinaro Technique is a bariactric surgery that proposes the stomach will be divide in two parts: a proximal part and a distal part for performing horizontal gastrectomy. Differently what will happen in the Modified Scopinaro Surgery that will divide the stomach in two parts: a proximal part and a distal part for performing gastroplasty.

SUMMARY:
The purpose of this study is to show that the modified technique Scopinaro surgery allows a better control or reduction of complications often found in nutritional pancreatic and biliary derivations, starting from the assumption of a modified technique is as effective as Scopinaro classical technique for reducing overweight and control of comorbidities in obese patients with grade II and III.

DETAILED DESCRIPTION:
28 participants Will be recruited and will be divided into 2 groups of 14 subjects each one. One group will receive the Classic Scopinaro surgery and the other, Modified Scopinaro Surgery. In Scopinaro Surgery Modified will be held with laparotomy and median opening in layers. It will also be performed at the manufacturing drifting pancreatic and biliary derivations, Roux-en-Y, dividing the small stomach.A communication portal to be implemented and calibrated through a nasogastric tube of 10mm where a retaining ring is placed horizontal gastroplasty, in order to avoid an expansion of this communication.

In the Classical Scopinaro surgery will be done the same procedures of Scopinaro Modified surgery , but the gastroplasty will be replaced by horizontal gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) > 35;
* Body Mass Index greater than or equal to 40;
* Be indicated for bariatric surgery after other attempts at treatment;
* If BMI > 35 and <40, must submit AT LEAST one of comorbidities below: Type II diabetes, dyslipidemia, hypertension, joint arthropathy in average or great, sleep apnea, hypothyroidism.

Exclusion Criteria:

* Pregnant or breastfeeding
* Had undergone bariatric surgery before.
* Diagnostic of psychiatric disorders, according to the evaluation of especialist.
* Be user of illegal drugs or alcohol abuse.
* Be severe disease carrier, according to an evaluation specialist.
* Have severe lung disease or liver cirrhosis, according to the evaluation of especialist.
* Being active virus carrier - HIV.
* Has any condition that prevents surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events | 18 months after the surgery.
  Patients will be followed for 18 months after surgery and will follow-up visits to collect information about body weight, complications from surgery, liver diseases, nutritional status, adverse events and evaluation of quality of life

SECONDARY OUTCOMES:
Number of patients that regain weight | 18 months after the surgery.
  Patients will be followed for 18 months after surgery and will follow-up visits to collect information about body weight.
deaths | 18 months from the surgery
  Number of patients that died

CONTACTS AND LOCATIONS:
Overall Officials: Paulo R Esselin de Melo, Principal Investigator — INSTITUTO PAULO REIS DE CLINICA CIRURGICA E OBESIDADE MORBIDA S/S
Locations (1):
- Instituto Paulo Reis de Clinica Cirurgica E Obesidade Morbida S/S, Goiânia, Goiás, Brazil